CLINICAL TRIAL: NCT04630626
Title: Extended Follow-up of Investigational Device Exemption (IDE) Subjects Treated With the Simplify Cervical Artificial Disc
Brief Title: Post-Approval Study Protocol for the Simplify Cervical Artificial Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P200022 PAS
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Degenerative Disc Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Simplify Disc (Experimental): Extended follow-up of IDE Subjects treated with the Simplify Cervical Artificial Disc during IDE G140154
  Interventions: Device: Simplify Disc
- Historical ACDF Control (Other): Historical ACDF Data from similar protocol used as control.
  Interventions: Other: ACDF

INTERVENTIONS:
Device: Simplify Disc — The Simplify Disc is a cervical artificial disc manufactured from polyether ether ketone (PEEK) endplates and a mobile, zirconia-toughened alumina ceramic core.
  Arms: Simplify Disc
Other: ACDF — Historical ACDF control data
  Arms: Historical ACDF Control

SUMMARY:
This study is intended to demonstrate the 5-year long-term safety and efficacy of the Simplify® Cervical Artificial Disc ("Simplify Disc") in subjects enrolled in the non-randomized Simplify Disc IDE study. This study was conducted under IDE G140154.

DETAILED DESCRIPTION:
This post approval study (PAS) is a continuation of the IDE pivotal study (G140154) as required under P200022. These data include long-term follow-up of subjects enrolled and treated under the IDE study from February 2016 to 2018 out to 60 months post-op. The control group is comprised of a historical ACDF population. Subjects were enrolled (signed consent) into the PAS on a rolling basis at either the 36 month, 48 month or 60 month visit based on their treatment date (under IDE G140154) and the date of PAS protocol approval. Data presented are compared to baseline data collected as part of the IDE study. Therefore, the start date and end dates of the PAS are not inclusive of the full 60 months of reported data.

ELIGIBILITY:
Inclusion Criteria:

- All subjects enrolled in the Simplify Disc IDE study are considered for this long-term follow-up study.

Exclusion Criteria:

* Subjects who were not implanted with the Simplify Disc during the IDE study
* Subjects who had a secondary surgical intervention at the index level during the IDE study
* Subjects who were withdrawn or withdrew consent to participate in the IDE study
* Subjects who do not consent to participate in long-term follow-up post-approval study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Orthopaedic Education and Research Institute of Southern California, Orange, California
  - USCD, San Diego, California
  - The Spine Institute for Spine Restoration, Santa Monica, California
  - Spine Education and Research Foundation, Thornton, Colorado
  - Kennedy-White orthopedic Center, Sarasota, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine institute of Louisiana, Shreveport, Louisiana
  - Rothman Institute, Egg Harbor, New Jersey
  - Buffalo Spine Surgery, Lockport, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Texas Spine Consultants, Addison, Texas
  - Texas Back Institute, Plano, Texas
  - Virginia Spine Institute, Reston, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No recruitment - long term follow up of subjects previously enrolled in IDE and historical control data
Period: Overall Study
Arm/Group | Simplify Disc | Historical ACDF Control
Started | 142 | 106 (Historical data)
Completed | 125 | 65 (Historical data)
Not Completed | 17 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simplify Disc | Historical ACDF Control | Total
Number analyzed (Participants) | 142 | 106 | 248
Age, Continuous [Median (Full Range); unit: years] | 43.2 [18.1 to 60.4] | 43.9 [27.8 to 59.3] | 43.6 [18.1 to 60.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 63 | 152
  Male | 53 | 43 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 123 | 93 | 216
  Black | 10 | 7 | 17
  Hispanic | 4 | 5 | 9
  Other | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142 | 106 | 248

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Composite Success, Parent IDE Study + Post Approval Study (PAS)
Description: Individual success for Simplify Disc and the historical control Anterior Cervical Discectomy and Fusion (ACDF) is defined as follows:
  * Improvement on the Neck Disability Index (NDI) of at least 15 percentage points compared to baseline in the Simplify Disc IDE study, and
  * No device failures by Month 60, and
  * No subsequent surgical procedure at the index level (including revision, removal, reoperation, or supplemental fixation) by Month 60.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 123 | 63
Participants | 117 | 40

2. Secondary Outcome: Number of Participants With Clinical Improvement in One or More Radicular Symptoms or Myelopathy (Neurological Status), Parent IDE Study + Post Approval Study (PAS)
Description: Endpoint includes the number of participates in each group that had improvement in one or more radicular symptoms or myelopathy based on their Neurological Status (motor exam, sensory exam, gait exam, and reflexes) at 60 months when compared to baseline data from the prior IDE study.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Population: Limited historical control neurological data available
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 122 | 23
Participants | 97 | 23

3. Secondary Outcome: Clinical Improvement in One or More Radicular Symptoms or Myelopathy (Visual Analog Scale), Parent IDE Study + Post Approval Study (PAS)
Description: Endpoint was examined using the Visual Analog Scale (VAS) for neck and arm pain which is a straight horizontal line of fixed length (100 millimeters) oriented from zero or no pain (best) to 100mm or the worst pain ever (worst).
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 124 | 65
score on a scale | 16.8 (12.1) | 23.8 (26.1)

4. Secondary Outcome: Participants Average Disc Height, Parent IDE Study + Post Approval Study (PAS)
Description: Disc height is calculated as a simple average of the anterior and posterior disc heights of the treated index level.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 121 | 63
mm | 4.06 (1.00) | 4.81 (1.17)

5. Secondary Outcome: Percentage of Participants With No Adjacent Level Disc Deterioration (ALDD) Superior Level, Parent IDE Study + Post Approval Study (PAS)
Description: Adjacent level disc deterioration looks at the quality of the disc space above (superior) and below (inferior) the treated index level on available radiographic images and each is graded as None, Mild, Moderate, Severe.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Population: Limited historical control data was available.
Measure: Number; unit: percentage of subjects with no ALDD
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 132 | 63
percentage of subjects with no ALDD | 52 | 6

6. Secondary Outcome: Percentage of Participants With No Adjacent Level Disc Deterioration (ALDD) Inferior Level, Parent IDE Study + Post Approval Study (PAS)
Description: as for outcome 5
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Population: Limited historical control data was available.
Measure: Number; unit: percentage of subjects with no ALDD
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 72 | 6
percentage of subjects with no ALDD | 59 | 10

7. Secondary Outcome: Percentage of Participants With No Displacement or Migration of the Device, Parent IDE Study + Post Approval Study (PAS)
Description: Displacement or Migration of the device will be compared device placement at 60 months to immediate post-op data collected under the IDE study (changes of >3 mm will be considered significant)
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Number; unit: percentage of subjects with no migration
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 122 | 60
percentage of subjects with no migration | 100 | 95

8. Secondary Outcome: Percentage of Participants Reporting Overall Treatment Satisfaction of "Very Satisfied" or "Satisfied", Parent IDE Study + Post Approval Study (PAS)
Description: Overall Treatment satisfaction was examined at 60 months. This was collected via a questionnaire completed by the subject. Response options to "How does the subject rate satisfaction with the treatment received?" included "Very Satisfied", "Satisfied", "Somewhat Satisfied", "Somewhat Dissatisfied", and "Very Dissatisfied". Response options to "If you could go back in time, would you choose to have the same treatment that you received for your neck condition?" included "Definitely Yes", "Probably Yes", "Maybe", "Probably Not" and "Definitely Not".
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Number; unit: % of "Very Satisfied"/"Definitely Yes"
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 125 | 63
% of "Very Satisfied"/"Definitely Yes"
  How does the subject rate satisfaction with the treatment recieved? | 83 | 75
  Would you choose to have the same treatment recieved? | 84 | 62

9. Secondary Outcome: Participants With Maintenance or Improvement on 12-Item Short Form Survey (SF-12), Parent IDE Study + Post Approval Study (PAS)
Description: 12-Item Short Form Survey (SF-12) is a questionnaire completed by the subject. Outcomes will be comparted at 60 months post treatment to baseline data collected from the IDE study.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Population: Questionnaire was only completed by subjects in the Simplify Disc arm. It was not collected for the historical control arm.
Measure: Number; unit: % of pts with maintenance or improvement
Arm/Group | Simplify Disc
Number analyzed (Participants) | 89
% of pts with maintenance or improvement
  Physical Component Score- PCS | 96
  Mental Component Score | 71.8

10. Secondary Outcome: Percentage of Participants With No Dysphagia Handicap Index (DHI), Parent IDE Study + Post Approval Study (PAS)
Description: Dysphagia Handicap Index (DHI) is a questionnaire completed by the subject. Outcomes at 60 months post-op were compared to baseline data collected under the IDE study.
Time Frame: IDE study 24 months + PAS 36 months = 60 months total
Measure: Number; unit: percentage of subjects with no Dysphagia
Arm/Group | Simplify Disc | Historical ACDF Control
Number analyzed (Participants) | 118 | 23
percentage of subjects with no Dysphagia | 97 | 100

ADVERSE EVENTS:
Time Frame: Data presented includes AEs collected under the Parent IDE study (G140154) and Post Approval Study (PAS). Data below represents AEs collected at post operative through 60 month follow up (IDE study 24 months + 36 months PAS)
Description: All adverse events were reviewed and adjudicated by an independent Clinical Events Committee.
Arm/Group | Simplify Disc | Historical ACDF Control
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/106
Serious Adverse Events (participants affected / at risk) | 25/132 | 17/106
Other Adverse Events (participants affected / at risk) | 105/132 | 72/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=132) | Historical ACDF Control (N=106)
Adjacent Segment Degeneration (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Gastrointestinal Complications (Gastrointestinal disorders) | 5 (5) | 1 (1)
Infection - Not At Surgical Site (Infections and infestations) | 3 (3) | 3 (4)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Trauma (General disorders) | 3 (3) | 1 (1)
Pain (Narcotic Given) (General disorders) | 1 (1) | 2 (2)
Surgery - Other Than the Spine (General disorders) | 2 (2) | 1 (2)
Radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Pain (No Narcotic Given) (General disorders) | 1 (1) | 2 (2)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ischemia (Vascular disorders) | 1 (1) | 1 (1)
Psychological Illness (Psychiatric disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Compressive Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Adverse Reaction or Allergy to Anesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infection at Surgical Site (Infections and infestations) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=132) | Historical ACDF Control (N=106)
Radiculopathy (Musculoskeletal and connective tissue disorders) | 37 (45) | 21 (30)
Spasm (Musculoskeletal and connective tissue disorders) | 33 (35) | 23 (34)
Inflammation Conditions (General disorders) | 23 (26) | 12 (15)
Adjacent Segment Degeneration (Musculoskeletal and connective tissue disorders) | 15 (18) | 10 (12)
Pain (No Narcotic Given) (General disorders) | 9 (9) | 16 (21)
Trauma (General disorders) | 20 (24) | 7 (9)
Pain (Narcotic Given) (General disorders) | 8 (8) | 19 (27)
Other (General disorders) | 15 (18) | 8 (10)
Infection - Not at Surgical Site (Infections and infestations) | 11 (13) | 4 (6)
Compressive Neuropathy (Nervous system disorders) | 8 (9) | 10 (11)
Headache (General disorders) | 8 (9) | 9 (11)
Increased Numbness (Nervous system disorders) | 12 (15) | 5 (8)
Gastrointestinal Complications (Gastrointestinal disorders) | 9 (10) | 0 (0)
Dysphagia (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (4)

LIMITATIONS AND CAVEATS:
Limited radiographic and neurological data for historical ACDF control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication results vary per investigator and per clinical trial agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04630626/Prot_SAP_000.pdf